CLINICAL TRIAL: NCT02010437
Title: A Randomised Clinical Trial Comparing Standard Cannula Delivered Foam Sclerotherapy, Catheter Directed Foam Sclerotherapy and ClariVein® Mechanochemical Ablation in the Management of Superficial Venous Insufficiency.
Brief Title: RCT Comparing Standard Cannula Delivered FS, UGFS and ClariVein® in the Management of SVI
Acronym: EVCA
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study design has been substantially revised and a new registration will be made in the future.
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: EVCA Trial
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Superficial Venous Insufficiency, Varicose Veins
Keywords: Superficial Venous Insufficiency
MeSH Terms: conditions — Varicose Veins | interventions — Sodium Tetradecyl Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Foam Sclerotherapy Group (Active Comparator): The axial vein will be cannulated under local anaesthesia and ultrasound guidance with the patient reclined in a supine position for GSV or ASV treatment, prone position if SSV or GV treatment.
  The foam is then prepared by the Tessari technique by the surgeon. Two 2-ml syringes will be connected via a three way stop-cock tap and a 5 micron filter in series (Braun Medical, Sheffield, UK). The syringes will contain 1 part Sodium Tetradecyl Sulphate 3% and 3 parts air. In practice 0.5ml of 3% STS will be drawn up against 2 ml of air. The foam will be produced by at least 20 passages from syringe to syringe through the filter.
  Up to 2ml of foam will be injected into each cannula under ultrasound control to observe venous spasm, followed by gentle massaging of the skin to propagate the foam through the segment of vein treated.
  Interventions: Drug: Sodium Tetradecyl Sulphate (STS)
- Catheter Directed Foam Sclerotherapy (CDS) Group (Active Comparator): The straight segment of axial vein will be cannulated under local anaesthesia at the lowest point of demonstrable reflux and a guide-wire inserted to facilitate the placement of the catheter system.The appropriate Unifuse® catheter will be selected and deployed through the introducer sheath and advanced to within 2cm of the junction or perforator at the upper limit of incompetence or the top of the incompetent segment in the case of segmental reflux. A 1:3 foam of 3% STD will be produced as described for FS. At this point the patient will be repositioned into a Trendelenburg position (head up)
  Interventions: Drug: Sodium Tetradecyl Sulphate (STS)
- ClariVein Group (CV) Treatment (Active Comparator): The straight segment of axial vein will be cannulated under local anaesthesia at the lowest point of demonstrable reflux and the ClariVein device 4-F micro sheath will be introduced up the vein via a guide wire as per manufacturer's instructions. Concentration of STD will depend on axial vein to be treated; if treating GSV or ASV 1.5% STD liquid will be used, if SSV or GV 1.0% STD liquid will be used. Volume of STD to be prepared for the CV treatment will be calculated using a dosage chart provided by the manufacturer
  Interventions: Drug: Sodium Tetradecyl Sulphate (STS)

INTERVENTIONS:
Drug: Sodium Tetradecyl Sulphate (STS)
  Other Names: Fibrovein

SUMMARY:
Leaking valves in the veins of the legs causes veins to become large and bloated. These swollen veins are called "varicose veins" and are a very common problem, affecting more than a third of all adults in the UK. Varicose veins reduce people's quality of life by causing problems such as pain, itching and restless legs. Varicose veins may also damage the skin over time causing problems such as bleeding, skin colour changes, eczema and even break-down in the skin which is called an ulcer. Newer, "key-hole" methods of treating leaky veins have been developed as an alternative to surgery and can be performed under local anaesthetic with the patient awake. Rather than cuts in the skin, these minimally invasive techniques are performed through tiny stab wounds; little larger than needle holes. The varicose vein is then destroyed from within, usually using heat to burn the inside of the vein. These procedures are popular; with a rapid recovery and a very high success rate. However these methods also require the vein to be surrounded by a large volume of dilute local anaesthetic which can to be slightly painful to administer. A technique called "Foam sclerotherapy" involves the injection of a drug which has been mixed into a foam. This goes into the vein and causes it to stick shut. This procedure is near painless to perform as very few, small local anaesthetic injections are required; however the chance for a successful treatment first time are lower and patients may need to return for repeat treatments to successfully treat the vein.

The aim of this study is to see whether the success rates for this technique can be improved. One method "catheter directed foam sclerotherapy" involves the delivery of the foam through a catheter (a long very thin tube), so that large lengths of vein can be treated through a single hole. The final method "ClariVein" again uses a catheter; but this time the catheter has a small wire on the end which spins around inside the vein; similar to an edge strimmer in the garden; except it irritates the vein: rather than cutting it. This irritation makes the vein more susceptible to the drug which can again be applied directly to the vein wall whilst it is still active. Early results show that this final method is very successful; however the equipment is more expensive than for the other two.

This study will randomly allocate willing participants with varicose veins to receive one of these three treatments to see whether the two newer treatments can improve the success rates and quality of life improvements seen with foam sclerotherapy, whilst also allowing near painless treatment, without significant complications, at an appropriate cost.

DETAILED DESCRIPTION:
. Investigational Plan Study Design This is a single centre three armed parallel group study with equal randomisation. The trial will be conducted in the Academic Vascular Surgical Unit of Hull York Medical School based at Hull Royal Infirmary, a university teaching hospital.

Target population The target population for this study are individuals with symptoms of SVI with ultrasound evidence of axial vein reflux and who have agreed to receive treatment for their axial vein reflux.

Recruitment Each patient referred to the vascular service with symptomatic SVI is assessed. Patients who potentially meet the inclusion criteria will be made aware of this research study and provided with the appropriate information, including the patient information sheet (see appendix 1). Patients will be given an opportunity to think about the invitation to participate and discuss with family/friends or other healthcare professionals if desired. Patients expressing an interest in participation will be offered an appointment for a screening visit with a study investigator.

Randomisation and Blinding Randomisation Participants will be randomised to one of the three treatments. Randomisation will be conducted by a sealed envelope system. Once enrolled in the study, efforts will be made to assess and manage all participants as outlined in the allocated treatment protocol until the pre-determined end-point of the study or until participant withdrawal. Following randomisation the participant's GP will be informed of the intended treatment modality Blinding Due to the nature of the procedures involved it will not be possible to blind the participant or clinical team as to which group the participant is allocated. Bias will be limited by the use of objective measurements, standardised protocols, use of patient reported outcomes and standardised assessor outcomes.

Power Calculation In order to detect a clinically significant difference in technical success of 15% with a power of 80% and a significance of 5%; 73 participants per group will be required. Assuming a 10% drop out rate we therefore aim to recruit 80 participants per group. The study will therefore randomise 240 participants in total over the 3 study groups.

Treatment Protocol All cases will be performed on a day-case, out-patient basis as per the standard practice in our unit by an experienced endovenous surgeon. For each participant, the investigating team will re-assess the inclusion and exclusion criteria, confirm the consent and undertake the procedure as per the protocol.

Participants judged to be at high risk of venous thromboembolic disease (VTE) due to the use of exogenous oestrogens, past medical history or a family history of VTE or thrombophilia or immobility will be given a single pre-operative dose of prophylactic molecular weight heparin (LMWH), in the absence of contraindications. All participants will have duplex assessment and marking using the same protocol with only the endovenous procedure differing.

The sclerotherapy drug used will be Sodium Tetradecyl Sulphate, also known as STD and marketed as Fibrovein® (STD Pharmaceutical Products, Hereford, UK). STD comes in different variations of concentration, for this trial we will use 3%, 1.5% or 1% STD depending on the procedure protocol. STD can be used as foam or as a liquid preparation which makes it ideal for our study. The STD used will be from routine stocks. It will be stored at room temperature in a suitably secure location in the ward, clinic or theatre. Careful records will be kept regarding which participants receive STD and its batch number Preoperative procedure The treatment aim is to eradicate any significant SVI present in the limb. Preoperatively the veins are marked by the surgeon using duplex-ultrasound with the patient standing. This will identify the extent and position of the refluxing axial vein alongside any incompetent perforating veins and varicose tributaries. The significant superficial varicose vein (GSV, ASV, SSV, GV) to be treated will have its length measured and noted. In addition, the average diameter of the varicose vein will be calculated via three transverse images of the vein (proximal, middle and distal) and noted. Potential areas to be punctured by cannulae may have local analgesia applied prior to treatment. The participant will be positioned supine on the operating table where in the Clarivein and Ultrasound Catheter group sterile precautions including disinfectant skin preparation and sterile draping will be employed, and the Foam Sclerotherapy and tributary treatment group skin disinfectant only. The ultrasound transducer will be prepared with a sterile covering and secured to the sterile drapes to allow sterile intra-operative ultrasound duplex scanning.

Operative Procedure: Foam Sclerotherapy Group The axial vein will be cannulated under local anaesthesia with an 18G (green), 20G (Pink) or 22G (Blue) Intravenous cannulae under ultrasound guidance with the patient reclined in a supine position for GSV or ASV treatment, prone position if SSV or GV treatment. This will be performed at the lowest point of demonstrable reflux and throughout the length of the incompetent vein at 20cm intervals. Each insufficient tributary system will also be cannulated separately. Venous blood will be aspirated and the cannulae flushed with normal saline to confirm that each is inside the target vein. Local anaesthesia can be used at each puncture site prior to needle insertion if desired by the patient. Once the cannulae are secured the leg is elevated to empty the veins.

The foam is then prepared by the Tessari technique by the surgeon. Two 2-ml syringes will be connected via a three way stop-cock tap and a 5 micron filter in series (Braun Medical, Sheffield, UK). The syringes will contain 1 part Sodium Tetradecyl Sulphate 3% and 3 parts air. In practice 0.5ml of 3% STS will be drawn up against 2 ml of air. The foam will be produced by at least 20 passages from syringe to syringe through the filter.

Up to 2ml of foam will be injected into each cannula under ultrasound control to observe venous spasm, followed by gentle massaging of the skin to propagate the foam through the segment of vein treated. The surgeon will also endeavour to prevent propagation of fresh foam beyond perforators and junctions into the deep venous system. The patient will be asked to dorsi-flex and plantar-flex their ankle several times to clear any foam which might have entered the deep venous system. At least 30 seconds will be left between each injection of foam. As per the European consensus guidelines a maximum of 12mls of foam will be used at one sitting32 33. Typical volumes of foam reported by Bradbury are 4-12ml in the GSV and 2-8 ml in the SSV34. After ensuring that the axial vein is treated the surgeon can then progress to the treating the tributaries and application of the dressings, as detailed below.

Operative Procedure: Catheter Directed Foam Sclerotherapy (CDS) Group The straight segment of axial vein will be cannulated under local anaesthesia at the lowest point of demonstrable reflux and a guide-wire inserted to facilitate the placement of the catheter system. The access cannulae will be removed and replaced with a 5F introducer sheath over a guide. A Unifuse® (AngioDynamics, Cambridge, UK) catheter system will be deployed via the sheath.

Unifuse® catheters available are 5F with either 45 cm or 90 cm lengths in combination with 5cm, 10cm or 15cm long infusion patterns. The appropriate Unifuse® catheter will be selected and deployed through the introducer sheath and advanced to within 2cm of the junction or perforator at the upper limit of incompetence or the top of the incompetent segment in the case of segmental reflux. The catheter will be aspirated to ensure correct position and flushed with normal saline. Each tributary system will be cannulated as was the case in the FS group.

A 1:3 foam of 3% STD will be produced as described for FS. At this point the patient will be repositioned into a Trendelenburg position (head up). The Unifuse® Self-Occluding ball wire will be inserted and the tip correctly positioned at 2cm from the junction under ultrasound guidance. As the internal diameter of the Unifuse® catheter is 1mm (3F) approximately 0.35ml of foam in the 45cm catheter or 0.7ml of form for the 90cm catheter will be injected to fill the dead-space. The appropriate volume of foam will be then be infused through the Unifuse® catheter during withdrawal under ultra-sound guidance. The catheter will be withdrawn the length of the infusion pattern following each injection. The surgeon will endeavour to prevent propagation of fresh foam beyond the perforators and junctions into the deep venous system. The maximum volume of foam used in one sitting is again limited to 12 ml, although the dead space in the catheter will be added to this. Once the varicose vein is treated the total volume of foam used is noted. After ensuring that the axial varicose vein is treated the surgeon can then progress to the treating the tributaries and application of the dressings, as detailed below.

Study Visits Baseline measurements will be collected from all participants once consent is obtained and prior to randomisation. Study measurements will be taken on the day of treatment and at the 1, 6, 12 and 52 week follow-up appointments, as detailed below Visit 1 (Baseline Assessment)

This assessment takes place after the signing of the consent form but prior to randomisation. Information collected will include:

* Identification and Demographic details

  o GP practice name with contact details
* Employment Status and Occupation

  o National Statistics Socio-economic Classification (NS-SEC)
* Medical History including

  * Previous investigations and treatments
  * Co-morbidities
  * Allergies and current medications
  * Mobility
* Clinical Examination including

  * Weight and Height
  * Venous Clinical Severity Score (VCSS)
  * CEAP Classification
* Photographic record of baseline limb appearance/bruising surface planimetry

  o Anterior, left lateral, posterior and right lateral aspects
* Duplex findings

  * Systems of insufficiency
  * Superficial Axis (GSV, AASV, SSV, Giacomini, non-axial)
  * Deep Axis
  * Perforators
* Quality of Life Measurements

  * EuroQol
  * SF-36 V2
  * AVVQ
  * CIVIQ Visit 2 (day of treatment) On the day of treatment the participant will undergo their randomised treatment as per the protocol. Technical and non-technical measurements will be recorded during this visit. Participants will also be given a 1-week Visual Analogue Diary and 1-week Analgesia Diary at this visit to be returned completed at visit 3 (1 week) Technical treatment measurements
* Vein axis/axes treated
* Number of tributary veins treated
* Length of axial vein and average diameter of vein
* Total duration of procedure

  * Duration of allocated procedure
  * Duration of tributary treatment
* Total volume of sclerotherapy (in ml) used per concentration

  * Volume of Sclerotherapy (in ml) delivered for allocated treatment
  * Volume of Sclerotherapy (in ml)delivered for tributary treatment
* Length and type of treatment catheter used (where applicable) Non-technical treatment measurements
* Visual analogue pain score (VAS)

  * During procedure (recorded immediately following the procedure)
  * Daily pain record for 1 week post procedure (recorded each evening in a patient diary)
* Daily analgesia diary for 1 week post procedure (with tablet numbers) Visit 3 (1 week post treatment) This visit should take place ±1 day from the target visit date.
* Collection of the 1 week VAS
* Collection of the 1 week Analgesia Diary
* Objective scoring of clinical severity. This will be assessed using both the VCSS and CEAP scores.
* Generic Quality of Life Assessments

  * EQ5D
  * SF36
  * SF6D
* Disease specific Quality of Life Assessments

  * AVVQ
  * CIVIQ
* The number, timing and nature of any further treatment required
* Satisfaction visual analogue scale
* Cosmesis visual analogue scale
* Bruising visual analogue scale
* Bruising surface planimetry
* Time to return to normal activities
* Number of primary care calls/visits related to this treatment
* Any additional secondary care costs related to this treatment (e.g. drugs to treat complications / additional clinic visits / days spent in hospital)
* Venous Duplex Ultrasound Visits 4, 5 and 6 (6, 12 and 52 weeks post treatment) These visits should take place ±7 day from the target visit date.
* Abbreviated medical history and clinical assessment
* Objective scoring of clinical severity. This will be assessed using both the VCSS and CEAP scores.
* Generic Quality of Life Assessments

  * EQ5D
  * SF36
  * SF6D
* Disease specific Quality of Life Assessments

  * AVVQ
  * CIVIQ
* Pain visual analogue scale
* Satisfaction visual analogue scale
* Cosmesis visual analogue scale
* Bruising visual analogue scale
* Bruising surface planimetry
* Time to return to normal activities
* Number of primary care calls/visits related to this treatment
* The number, timing and nature of any further treatment required
* Any additional secondary care costs related to this treatment (e.g. drugs to treat complications / additional clinic visits / days spent in hospital)
* Venous Duplex Ultrasound Additional Treatment Visits Participants who undergo additional treatments (as per treatment protocol) will require an additional "baseline" and set of measurements as detailed below. Visits will be identified with the prefix A, B, C… etc. to differentiate between treatment rounds if more than one session is required.

Visit A0 (Additional Treatment Baseline)

* Objective scoring of clinical severity. This will be assessed using both the VCSS and CEAP scores.
* Generic Quality of Life Assessments

  * EQ5D
  * SF36
  * SF6D
* Disease specific Quality of Life Assessments

  * AVVQ
  * CIVIQ
* Photographic record of baseline limb appearance

  o Anterior, left lateral, posterior and right lateral aspects
* Duplex findings

  * Systems of insufficiency
  * Superficial Axis (GSV, AASV, SSV, Giacomini, non-axial)
  * Deep Axis
  * Perforators Visit A2 (Retreatment Visit) On the day of treatment the participant will undergo their original randomised treatment as per the protocol unless the participant requests a different treatment or the responsible clinician feels that this is not in the patient's interest. If symptoms are related to incompetent tributaries, the tributary varicose vein treatment protocol will be used for treatment. Technical and non-technical measurements will be recorded. Participants will again also be given a 1-week Visual Analogue Diary and 1-week Analgesia Diary at this visit to be returned at visit A3 (1 week) Technical treatment measurements
* Vein axis/axes treated
* Number of tributary veins treated
* Length of axial vein and average diameter of vein
* Total duration of procedure

  * Duration of allocated procedure
  * Duration of tributary treatment
* Total volume of sclerotherapy (in ml) used per concentration

  * Volume of Sclerotherapy (in ml) delivered for allocated treatment
  * Volume of Sclerotherapy (in ml)delivered for tributary treatment
* Length and type of treatment catheter used (where applicable) Non-technical treatment measurements
* Visual analogue pain score (VAS)

  * During procedure (recorded immediately following the procedure)
  * Daily pain record for 1 week post procedure (recorded each evening in a patient diary)
* Daily analgesia diary for 1 week post procedure Visit A3 (1 week post retreatment) This visit should take place ±1 day from the target visit date.
* Collection of the 1 week VAS
* Collection of the 1 week Analgesia Diary
* Objective scoring of clinical severity. This will be assessed using both the VCSS and CEAP scores.
* Generic Quality of Life Assessments

  * EQ5D
  * SF36
  * SF6D
* Disease specific Quality of Life Assessments

  * AVVQ
  * CIVIQ
* Visual analogue satisfaction scale
* Visual analogue cosmesis scale
* Visual analogue bruising scale
* Bruising surface planimetry
* Time to return to normal activities
* Number of primary care calls/visits related to this treatment
* Any additional secondary care costs related to this treatment (e.g. drugs to treat complications / additional clinic visits / days spent in hospital)
* Venous Duplex Ultrasound After this visit the participant will be followed up at the next scheduled routine appointment.

The primary outcome of this trial is the technical success rate of treatment at 1 year. The ultrasound appearances of the axial vein will be categorised as:

* Fully occluded
* Partial recanalisation (≤15% by length)
* Widespread recanalisation (>15% by length). Secondary Outcomes Procedural - technical
* Vein axis/axes treated
* Number of tributary veins treated
* Length of axial vein and average diameter of vein
* Total duration of procedure

  * Duration of allocated procedure
  * Duration of tributary treatment
* Total volume of sclerotherapy (in ml) used per concentration

  * Volume of Sclerotherapy (in ml) delivered for allocated treatment
  * Volume of Sclerotherapy (in ml)delivered for tributary treatment
* Length and type of treatment catheter used (where applicable) Post procedure
* Subjective treatment pain

  * during the procedure
  * 1 week post procedure
* Analgesia requirements for 1 week per treatment
* Time to return to normal activities.
* Subjective bruising assessment
* Subjective satisfaction
* Subjective cosmetic change
* Objective bruising assessment
* Change in clinical severity

  * VCSS
  * CEAP.
* Change in generic Quality of Life

  * EQ5D
  * SF36
  * SF6D
* Change in disease specific Quality of Life

  * AVVQ
  * CIVIQ
* The number, timing and nature of any further treatment required
* Total number of primary care calls/visits related to this treatment
* Any additional secondary care costs related to this treatment
* Duplex Ultrasound measurements (proximal, middle and distal vein diameter) Expected Value of results Our proposed project would be the first to compare these three tumescent-free endovenous-ablative techniques. This will provide patients with a greater choice in their treatment and will usher in the next logical stage in endovenous treatments

ELIGIBILITY:
Inclusion Criteria:

* • Aged 18 or over

  * Symptomatic superficial venous insufficiency; Clinical grades C2 - C6; which will likely benefit from treatment in the opinion of an experienced specialist and the participant
  * Superficial axial incompetence with proposed treatment lengths of >10cm. This axis may be a great saphenous vein (GSV), anterior accessory saphenous vein (ASV), small saphenous vein (SSV) or Giacomini vein (GV). Multiple veins can be treated.
  * The proposed treatment length is straight enough to be cannulated with the catheter devices and the SVI is suitable for treatment with any modality in the study in the view of an experienced specialist
  * Willing to participate (including acceptance of randomisation to either treatment) and give valid, informed consent

Exclusion Criteria:

* • Inability to give informed written consent

  * Unsuitable for any of the treatments in the opinion of a suitably experienced specialist.
  * Unwilling or inability to comply with the requirements for follow-up visits.
  * Known allergy to any of the key medications used in the treatment protocols
  * Known right to left circulatory shunt
  * Evidence of deep venous thrombosis or occlusion
  * Active or recent thrombophlebitis (within 6 weeks)
  * Impalpable foot pulses and an Ankle-Brachial Pressure Index of less than 0.8
  * Pregnancy
  * Active malignancy
  * Immobility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
technical success rate of treatment at 1 year | 1 year
  The primary outcome of this trial is the technical success rate of treatment at 1 year. The ultrasound appearances of the axial vein will be categorised as:
  * Fully occluded
  * Partial recanalisation (≤15% by length)
  * Widespread recanalisation (>15% by length).

SECONDARY OUTCOMES:
Disease Specific Quality of Life (Aberdeen Varicose Vein Questionnaire AVVQ) | 1 Year
  The Aberdeen Varicose Vein Questionnaire (AVVQ) is a disease specific Quality of Life questionnaire which measures the QoL impairment associated with venous disease42. It is one of the most widely used venous disease specific QoL measurements and has been extensively validated43. The AVVQ consists 14 multiple choice questions and an unmarked diagram of the front and rear aspects of a pair of legs. The subject is invited to draw the distribution of their varicose veins on this diagram and the assessor uses a standardised acetate overlay with a grid pattern to score the number of affected segments. The AVVQ result has the added benefit over generic questionnaires in that it is more sensitive to small but significant differences in the health state of people with venous disease

CONTACTS AND LOCATIONS:
Locations (1):
- Hull Royal Infirmary, Hull, United Kingdom